CLINICAL TRIAL: NCT04753385
Title: The RECOVER sUb-study, Which Leverages quaNtitative and Credible Research tOols From Verily, Will providE Assessment measuRes for Depressive Episodes
Acronym: UNCOVER
Status: Terminated | Type: Observational
Why Stopped: UNCOVER terminated early based on low enrollment and lack of device data collected making analysis unfeasible.
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: LND300
Record Dates: First submitted 2021-01-07; First posted 2021-02-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; TRD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect both active and passive data using a wearable, multi-sensor device (Verily Study Watch) and phone application (Mood App) which aims to capture mental health status, in subjects participating in the RECOVER clinical trial (A Prospective, Multi-center, Randomized Controlled Blinded Trial Demonstrating the Safety and Effectiveness of VNS Therapy® System as Adjunctive Therapy Versus a No Stimulation Control in Subjects With Treatment-Resistant Depression).

DETAILED DESCRIPTION:
A prospective, observational, exploratory study collecting passive and active behavioral, environmental and physiological data, via the use of an Android smartphone application and Study Watch.

This sub-study is only open to sites participating in the RECOVER clinical study.

All subjects participating in the RECOVER clinical trial at active UNCOVER sites will be offered participation in this sub-study.

Subjects who opt-in to the Mood App portion of the sub-study will be followed for a minimum of 12 months and a maximum of 60 months for the Mood App portion of the sub-study.

Subjects who opt-in to the use of the Study Watch portion of the sub-study will be followed for a minimum of 12 months and maximum of 24 months for the Study Watch portion of the sub-study.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

1. Current consented subject in the RECOVER clinical trial;
2. Adult (i.e. ≥ 18 years of age, unless a resident of any U.S. state where the age of majority is 19, in which case must be ≥ 19 years of age);
3. Able and willing to provide written informed consent for this sub-study;
4. Able and willing to comply with all study procedures;
5. Able to read and speak English.

Phone Application

1. Have a personal Google user account or be willing to create and own a personal Google user account;
2. Owns a personal Android smartphone with a data plan and is the sole user of that smartphone;
3. Agrees to download and maintain the phone application onto personal Android smartphone for the duration of the sub-study;

Study Watch

1. Willing to comply with Study Watch wearing and recharging requirements

Exclusion Criteria:

All Subjects

1. Any condition or situation the Principal Investigator determines as inappropriate for study inclusion

Phone Application

No additional exclusion criteria for phone application

Study Watch

1. Subjects with known severe allergy to nickel or metal jewelry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This sub-study is only open to sites participating in the RECOVER clinical study.
  All subjects participating in the RECOVER clinical trial at active UNCOVER sites will be offered participation in this sub-study.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Percentage of PHQ-8 tasks | Through study completion; Average 2 years
  Percentage of PHQ-8 tasks completed over the duration of the study
Percentage of Voice Diary tasks | Through study completion; Average 2 years
  Percentage of Voice Diary tasks completed over the duration of the study
Number of ping sensor recordings | Through study completion; Average 2 years
  Number of ping sensor recordings over the duration of the study
Number of hours of watch wear time | Through study completion; Average 2 years
  Number of hours of watch wear time over the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Charles Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Keck Hospital of USC, Los Angeles, California
  - SF-Care, Inc., San Rafael, California
  - Kind Research Group, Boca Raton, Florida
  - APG Research, LLC, Orlando, Florida
  - Nova Psychiatry Inc., Orlando, Florida
  - Advanced Mental Health Care Inc., Royal Palm Beach, Florida
  - Florida Center for TMS, Saint Augustine, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - AMR-Baber Research, Inc., Naperville, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Beacon Medical Group Behavioral Health, South Bend, Indiana
  - Sheppard Pratt Health Systems, Baltimore, Maryland
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Psychiatric Care and Research, O'Fallon, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Hapworth Research Inc., New York, New York
  - Center for Neuropsychiatry and Brain Stimulation (CNBS), Cary, North Carolina
  - Ohio State University, Columbus, Ohio
  - OU-SOCM Dept of Psychiatry, Tulsa, Oklahoma
  - Scranton Medical Institutes, Moosic, Pennsylvania
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - UT Health Austin, Austin, Texas
  - UT Center of Excellence on Mood Disorders, Houston, Texas
  - North Pointe Psychiatry, Lewisville, Texas
  - Neuropsychiatric Associates, Plc, Woodstock, Vermont
  - Carilion Clinic, Roanoke, Virginia
  - Seattle Neuropsychiatric Treatment Center, Bellevue, Washington
  - Center for Anxiety and Depression, Mercer Island, Washington